CLINICAL TRIAL: NCT04847024
Title: Parecoxib vs. Dexketoprofen in Combination With Acetaminophen as Additional Analgesia in Patients With Neuraxial Morphine for the Management of Pain After Cesarean Section. A Randomized, Double Blind, Controlled Trial.
Brief Title: Parecoxib vs. Dexketoprofen for the Management of Pain After Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-523
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Caesarean Section; Pain
Keywords: Caesarean section; Pain; Parecoxib; Dexketoprofen
MeSH Terms: conditions — Pain | interventions — parecoxib; dexketoprofen trometamol

STUDY DESIGN:
Intervention Model Description: Parecoxib + acetaminophen vs Dexketoprofen + acetaminophen in patient receiving neuraxial analgesia for pain after caesarean section.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parecoxib (Experimental): Parecoxib 40 mg reconstituted in 2ml of saline solution, to pass IV as a bolus, every 12hrs + acetaminophen 1g in 100cc of saline solution to pass IV in 15 minutes, every 6hrs.
  Interventions: Drug: Parecoxib
- Dexketoprofen (Experimental): Dexketoprofen 50 mg in 100 cc of saline solution, protected from sunlight, to be given IV in 15 minutes, every 8hrs + acetaminophen 1g in 100 cc of saline solution to be given IV in 15 minutes, every 6hrs.
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Parecoxib — 40 mg IV
  Arms: Parecoxib
Drug: Dexketoprofen — 50 mg IV
  Arms: Dexketoprofen

SUMMARY:
Although it is known that parecoxib and dexketoprofen are commonly used in successful post-operative pain relief, there are very few studies that compare these two agents in their individual applications and/or combined with neuraxial analgesia with opioids and even less in post-cesarean section pain, as well as the evaluation of the side effects and their impact on the patient's functionality. For this reason, in order to approach this answer, we sought to perform this study in patients undergoing elective or emergency cesarean section in our institution, who meet the inclusion criteria, using the Visual Analog Pain Scale at 12 hrs and 24 hrs post surgery and evaluating the aforementioned side effects, comparing in one arm of the study Parecoxib + acetaminophen vs Dexketoprofen + acetaminophen in the other arm, randomizing the patients in both groups using a double-blind configuration.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy 32w or more.
* Emergency or elective caesarean section.

Exclusion Criteria:

* Allergy to Parecoxib.
* Allergy to dexketoprofen.
* Allergy to acetaminophen.
* General anesthesia.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gender identity
Enrollment: 380 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Pain at 12 hours | 12 hours
  Evaluation of pain using the Visual Analogue Scale (from 0 to 10, where 0 is no pain and 10 is the most terrible pain imaginable)
Pain at 24 hours | 24 hours
  Evaluation of pain using the Visual Analogue Scale (from 0 to 10, where 0 is no pain and 10 is the most terrible pain imaginable)

SECONDARY OUTCOMES:
Side effects | 24 hours
  Side effects associated with the drug used (Dexketoprofen vs. Parecoxib)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No